CLINICAL TRIAL: NCT03704545
Title: Clinical Impact of Pharmaceutical Consultations in Patients Treated for Chronic Obstructive Pulmonary Disease at Home
Acronym: BPCObs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2017-03/JMK-01; 2018-A01699-46 (Other: ANSM)
Record Dates: First submitted 2018-10-10; First posted 2018-10-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2023-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention)
- Experimental group from the hospital (Experimental)
  Interventions: Other: Pharmaceutical consultation at the hospital
- Experimental group from the city (Experimental)
  Interventions: Other: Pharmaceutical consultation at the pharmacy; Other: Follow-up pharmaceutical consultation at the pharmacy

INTERVENTIONS:
Other: Pharmaceutical consultation at the hospital — During 20 minutes, the patient will be educated about chronic obstructive pulmonary disease treatments and their use.
  Arms: Experimental group from the hospital
Other: Pharmaceutical consultation at the pharmacy — During 20 minutes, the patient will be educated about chronic obstructive pulmonary disease treatments and their use.
  Arms: Experimental group from the city
Other: Follow-up pharmaceutical consultation at the pharmacy — During 10 minutes, the patient will get more information about his chronic obstructive pulmonary disease treatments and their use.
  Arms: Experimental group from the city

SUMMARY:
The implementation of pharmaceutical consultations in the city or at the hospital could modify the occurrence of exacerbations related to chronic obstructive pulmonary disease after return of the patient to his home.

ELIGIBILITY:
Inclusion Criteria:

* The patient has signed the consent form.
* The patient is affiliated to a health insurance programme
* The patient is at least 18 years old (≥).
* The patient is admitted to complete hospitalization (for patients in the "Hospital and Control" groups).
* The patient is diagnosed with stage 2 to 4 Chronic Obstructive Pulmonary Disease. The diagnosis as well as the stage of the disease are validated by a pulmonologist at the facility.
* The patient has one or more inhaler devices to treat Chronic Obstructive Pulmonary Disease.
* The patient returns to his / her home when discharged from hospital (for patients in the "Hospital and Control" groups).
* The patient is available for a follow-up of 12 months.

Exclusion Criteria:

* The subject participates in another interventional study.
* The subject is in an exclusion period determined by a previous study.
* The patient is under safeguard of justice.
* The subject refuses to sign the consent.
* It is not possible to give the patient (or his/her trusted-person) informed information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Number of exacerbation events | Month 3
  Exacerbation events will be defined as any episode of increased respiratory symptoms, especially dyspnea, cough and sputum production, and increased sputum purulence.
Number of exacerbation events | Month 6
  Exacerbation events will be defined as any episode of increased respiratory symptoms, especially dyspnea, cough and sputum production, and increased sputum purulence.
Number of exacerbation events | Month 9
  Exacerbation events will be defined as any episode of increased respiratory symptoms, especially dyspnea, cough and sputum production, and increased sputum purulence.
Number of exacerbation events | Month 12
  Exacerbation events will be defined as any episode of increased respiratory symptoms, especially dyspnea, cough and sputum production, and increased sputum purulence.

SECONDARY OUTCOMES:
Number of visits to the attending physician | Month 3
Number of visits to the attending physician | Month 6
Number of visits to the attending physician | Month 9
Number of visits to the attending physician | Month 12
Number of visits to the pulmonologist | Month 3
Number of visits to the pulmonologist | Month 6
Number of visits to the pulmonologist | Month 9
Number of visits to the pulmonologist | Month 12
Number of visits to the hospital emergency service | Month 3
Number of visits to the hospital emergency service | Month 6
Number of visits to the hospital emergency service | Month 9
Number of visits to the hospital emergency service | Month 12
Number of hospitalisation events | Month 3
Number of hospitalisation events | Month 6
Number of hospitalisation events | Month 9
Number of hospitalisation events | Month 12
Medication Possession Ratio | 12 months
  unit = percent
Usability score of devices | Month 3
  Score between 0 and 3
Usability score of devices | Month 6
  Score between 0 and 3
Usability score of devices | Month 9
  Score between 0 and 3
Usability score of devices | Month 12
  Score between 0 and 3
Quality of life questionnaire | Month 1
  The quality of life questionnaire BPCO-VQ11 is composed of 11 items. Each item is scored in a 5 point scale.
Quality of life questionnaire | Month 6
  The quality of life questionnaire BPCO-VQ11 is composed of 11 items. Each item is scored in a 5 point scale.
Quality of life questionnaire | Month 12
  The quality of life questionnaire BPCO-VQ11 is composed with11 items. Each item is scored in a 5 point scale.
device usage learning curve | 12 months
satisfaction questionnaire | Month 12
  This questionnaire is composed with 4 questions. Each item is scored in a 4 point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Nimes University Hospital, Nîmes, France

REFERENCES:
- [Result] Hachemi D, Leguelinel-Blache G, Bouvet S, Roux-Marson C, Plouvier N, Kinowski JM, Castelli C, Dubois F. Clinical impact of pharmaceutical consultations in patients treated for chronic obstructive pulmonary disease: Study protocol for a randomized controlled trial (BPCObs study). Contemp Clin Trials Commun. 2023 Dec 20;37:101249. doi: 10.1016/j.conctc.2023.101249. eCollection 2024 Feb. PMID 38269046